CLINICAL TRIAL: NCT01292980
Title: Air Fluidized Therapy Use in Patients Who Present With Suspected Deep Tissue Injury - a Case Series
Brief Title: Air Fluidized Therapy (AFT) in Patients With Suspected Deep Tissue Injury (sDTI)
Status: Completed | Type: Observational
Sponsor: Hill-Rom (Industry)
Responsible Party: Catherine VanGilder, Hill-Rom
Other Study IDs: CR-2009-08
Record Dates: First submitted 2011-02-08; First posted 2011-02-10 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Pressure Ulcers
Keywords: sDTI; Pressure ulcers; Therapy surfaces; Mattresses; Deep Tissue Injury; pressure ulcer treatment
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: AFT bed — All identified patients will receive a AFT bed for a maximum of 21 days or until discharge
  Other Names: Clinitron® Rite HiteTM bed

SUMMARY:
Patients with a suspected Deep Tissue Injury (or a purple reddened area over a bony prominence of their body, which is expected to break down into a pressure ulcer) will be place on the Clinitron® Rite HiteTM bed to see if the air fluidized mattress decreases the amount of tissue breakdown from their bruise.

DETAILED DESCRIPTION:
Up to 15 centers will participate in this case series in acute care and long term acute care facilities. Patients who present with sDTI and consent for study will have the Clinitron® Rite HiteTM bed ordered and delivered within a 12 hour window to be able to participate. They will have their sDTI photographed, and an assessment of expected breakdown will be noted by the clinical team. The patient will be followed during the course of hospitalization and additional photographs and documentation will be performed by the clinical team to demonstrate the actual breakdown that occurred.

Information including the pertinent history of current illness, co-morbid conditions, and demographic information will be shared with the sponsor in order to demonstrate each case.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with sDTI on the supine aspect of their body
2. Patient does not require a pulmonary specialty bed for care
3. Patient is expected to be in the hospital for at least 3 days
4. Patient weighs between 30 and 350 Lbs.
5. Patient's height is less than 75 inches tall
6. Patient, or patient's representative, is willing and able to sign written informed consent
7. Patient is expected to survive hospitalization.

Exclusion Criteria:

1. Patient is less than 18 years of age
2. Patient has already participated in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who present to the hospital with SDTI
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2010-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Degree of breakdown | 21 days
  This case series seeks to identify patients with suspected DTI and capture actual patient outcomes with AFT treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Harris Methodist Hospital, Fort Worth, Texas, United States